CLINICAL TRIAL: NCT07036432
Title: Introduction of EndoSign ® in Management of Barrett's Oesophagus - a Swedish Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIV-23-06-043373
Record Dates: First submitted 2025-06-02; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Barrett Esophagus
Keywords: endosign; capsule sponge
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endosign (Other)
  Interventions: Device: Endosign

INTERVENTIONS:
Device: Endosign — The intervention involves the EndoSign® Cell collection device (Cyted Ltd), a non-endoscopic method for esophageal sampling.
  Patients swallow a gelatine/HPMC capsule containing a sponge attached to a string. After ~7 minutes in the stomach for dissolution and sponge expansion, a trained nurse withdraws the sponge via the string, collecting cells. Optional throat anesthetic is offered.
  It can be performed without sedation in an outpatient clinic setting by a nurse. Samples undergo central analysis for TFF3, atypia, and p53, differing from standard biopsy histopathology. This study specifically evaluates its feasibility, acceptability, and nurse-led implementation in Swedish hospitals for Barrett's surveillance.

SUMMARY:
This study is looking at a new way to detect and monitor Barrett's esophagus (BE), a condition where the lining of the esophagus changes, increasing the risk of esophageal cancer. Currently, monitoring involves an endoscopy, where a camera is passed down the throat. While effective, endoscopy can be uncomfortable, uses significant healthcare resources, and sometimes involves sedation.

This Swedish study explores a less invasive method called EndoSign®. EndoSign® is a small, swallowable capsule containing a sponge attached to a thin string. Patients swallow the capsule with water. It dissolves in the stomach over about 7 minutes, releasing the sponge. A trained nurse then gently pulls the sponge back up through the esophagus using the string, collecting cells along the way. The whole visit takes about 20-30 minutes. These cells are then sent to a lab to be checked for signs of BE and early changes (like TFF3, atypia, and p53) that might indicate a higher risk.

The main goals of this study are:

To see if using EndoSign® is practical (feasible) in several Swedish hospitals.

To find out how patients feel about the EndoSign® test - is it acceptable and comfortable?.

To check how safe the EndoSign® procedure is.

To gather information needed to plan larger studies in the future.

Who is participating? Around 70 adults (aged 18-84) across five Swedish hospitals, who have a confirmed diagnosis of BE and are already part of a surveillance program, are enrolled. Patients with certain alarm symptoms or those scheduled for immediate treatment are excluded.

What happens in the study? Participants have a separate visit for the EndoSign® test, performed by a trained nurse. They also undergo their regular surveillance endoscopy (at least 90 days after the capsule test). Participants fill out questionnaires about their experience, comfort, and preferences after both procedures and again at 7 and 90 days.

Potential Benefits & Risks:

EndoSign® could offer a simpler, less invasive, and potentially more comfortable way to monitor BE, which might reduce the need for some endoscopies. Early results show it is well-tolerated, with most patients preferring it over endoscopy, and has a high success rate and safety profile. Risks are low, with the most common being a temporary sore throat. Serious complications are considered very rare.

This feasibility study aims to provide evidence on whether EndoSign® can be a valuable addition to BE surveillance in Sweden, potentially improving patient experience and resource use.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histopathologically confirmed diagnosis of Barrett's esophagus, specifically showing intestinal metaplasia.
* Patients must have at least a C0M1 Prague classification for their Barrett's esophagus.
* Patients must be under active monitoring with a surveillance endoscopy already planned to occur within the next 3 to 12 months.
* Patients must be between 18 and 84 years of age.

Exclusion Criteria:

* Patients scheduled for any endoscopic treatment (such as ablation) during their upcoming surveillance endoscopy.
* Patients experiencing alarm symptoms, including:
* Dysphagia (difficulty swallowing) and/or food sticking.
* Dyspepsia (indigestion) combined with weight loss.
* Dyspepsia combined with anaemia.
* Patients with a current diagnosis of an oropharyngeal, esophageal, or gastro-oesophageal tumour.
* Patients who have received treatment to their esophagus (e.g., endoscopic mucosal resection (EMR), endoscopic submucosal dissection (ESD), radiofrequency ablation (RFA), or surgery) within the last two months.
* Patients known to have gastric or oesophageal varices or cirrhosis of the liver.
* Patients with any known anomaly of the oesophagus, such as webbing, pouches, or strictures.
* Patients who are unable to provide informed consent.
* Patients who have had a stroke or possess any other neurological disorder that has affected their swallowing ability.
* Patients who have experienced a myocardial infarction (heart attack) within the past 3 months.
* Patients who have undergone fundoplication or any other surgery involving the esophagus and proximal (upper) stomach.
* Patients currently using anti-trombotic medications which cannot be safely stopped temporarily for the procedure.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Technical Success Rate of the EndoSign® Procedure | Perioperative/Periprocedural
  Measures the rate of successfully completed EndoSign® procedures. Technical success is defined as a participant successfully swallowing the capsule (in a maximum of two attempts) and subsequent successful retrieval of the sponge by the nurse.
Patient-Reported Acceptability and Experience of the EndoSign® Procedure Compared to Gastroscopy | Perioperative/Periprocedural and at 7 and 90-day follow-ups. (Both Visits)
  Measures and compares patient-reported outcomes for both the EndoSign® procedure and the surveillance gastroscopy. This includes Visual Analog Scale (VAS) scores (0-10) for discomfort and pain, which are measured immediately post-procedure and 15 minutes later for each respective procedure. It also assesses the patient's willingness to undergo each procedure again and their stated preference for future surveillance.
  Patient willingness to undergo the EndoSign® procedure again. Patient preference for EndoSign® vs. endoscopy for future surveillance.
Safety of the EndoSign® Procedure | Perioperative/Periprocedural and up to 90 days post-procedure.
  Incidence and rates of all Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Serious Adverse Device Effects (SADEs) are recorded following the EndoSign® procedure. Events are classified by severity and relatedness.

SECONDARY OUTCOMES:
Sample Adequacy of the EndoSign® Procedure | Perioperative/Periprocedural
  The proportion of retrieved EndoSign® samples are deemed adequate for full laboratory analysis, including TFF3 expression, atypia assessment, and p53 immunohistochemistry. An inadequate sample may be due to insufficient columnar cells or other factors preventing full analysis.
Risk Stratification Performance of the EndoSign® Test | Perioperative/Periprocedural
  Evaluation of the EndoSign® test's ability (using TFF3, atypia, p53, and clinical factors) to classify patients into low, moderate, and high-risk groups for harboring dysplasia. This includes calculating metrics such as Negative Predictive Value (NPV) for no dysplasia in low/moderate-risk groups and Positive Predictive Value (PPV) for dysplasia in the high-risk group, by comparing with endoscopic biopsy findings.
Assessment of Patient-Reported Health-Related Quality of Life using EQ-5D-5L | Perioperative/Periprocedural and at 7 and 90-day follow-ups.
  Measurement of general health-related quality of life using the EQ-5D-5L questionnaire, which assesses five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and includes a self-rated health Visual Analog Scale (VAS).
EndoSign® Capsule Swallowing Attempts | Perioperative/Periprocedural
  The number of attempts required for patients to successfully swallow the EndoSign® capsule. Swallowing success contributes to the overall technical feasibility.

OTHER OUTCOMES:
Mean Cost per procedure for Implementation of the EndoSign® Procedure | Through study completion, average 8 months
  The total cost of implementation, including materials (EndoSign® kit, sampling materials), staff time, and laboratory analysis (TFF3), is divided by the total number of completed procedures. The result is reported in SEK per procedure.
Mean Number of Supervised Procedures Required for a Healthcare Professional to Achieve Competency. | Perioperative/Periprocedural
  Mean number of EndoSign® procedures a nurse needs to perform under supervision before being deemed competent for independent practice.
Clinical Staff Acceptability of the EndoSign® Procedure Experience | At the end of the recruitment period at each individual study site.
  Staff experience and acceptability is evaluated using a structured survey that includes both Likert scales and open-ended questions. The survey covers key domains such as the nurses' training, procedural experience, and implementation perspectives.
Mean Turnaround Time for Laboratory Analysis of EndoSign® Samples. | Throughout the study's active procedural and analysis phase.
  Measures the number of calendar days from the time a sample is sent from the hospital site to the laboratory in the UK until the test result is received
Feasibility of Patient Recruitment | Baseline (during screening)
  To assess the feasibility of recruitment by determining the proportion of eligible patients who consent to participate out of the total number of patients invited. This also includes quantifying the number of patients potentially available for recruitment from surveillance programs at each site. Recruitment feasibility is tracked via screening logs.
Evaluation of Data Collection Methods and Outcome Measure Completeness | From baseline (Visit 1) through all patient follow-up points (up to 90 days post-gastroscopy for the final patient)
  To evaluate the feasibility of the data collection methods, including response rates for questionnaires (e.g., VAS, preference questionnaires, EQ-5D) at baseline and follow-ups. This also includes tracking withdrawal and drop-out rates, and follow-up completion rates.
Descriptive Comparison of EndoSign® Biomarker Findings with Matched Endoscopic Biopsy Histopathology | Perioperative/Periprocedural
  A descriptive analysis comparing the EndoSign® test results (TFF3 status, presence/absence of atypia, p53 expression status) with the histopathological findings from the patient's subsequent surveillance endoscopy biopsies (e.g., presence/absence of intestinal metaplasia, grade of dysplasia).

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - Vrinnevi Hospital, Norrköping
  - Ersta Hospital, Stockholm
  - Karolinska University Hospital, Stockholm

DOCUMENTS (1):
  • Study Protocol (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT07036432/Prot_000.pdf